CLINICAL TRIAL: NCT00447967
Title: A Randomized Phase II Study of Irinotecan and Oxaliplatin Versus the Combination of 5-FU/LV and Oxaliplatin, as First-Line Treatment in Patients With Locally Advanced or Metastatic Gastric Cancer
Brief Title: Combination of CPT-11 and LoHP vs Combination of 5-FU, Leucovorin and LoHP as 1st Line Treatment in Gastric Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: I.Boukovinas, Hellenic Oncology Research Group
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/04.18
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Gastric Cancer
Keywords: Metastatic Gastric Cancer; Oxaliplatin; Irinotecan
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): IOX
  Interventions: Drug: Irinotecan; Drug: Oxaliplatin
- 2 (Experimental): FLOX
  Interventions: Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 200 mg/m2 IV on Day 1 every 3 weeks for 6 cycles
  Other Names: CPT-11
  Arms: 1
Drug: Oxaliplatin — Oxaliplatin 80 mg/m2 IV on Day 2 every 3 weeks for 6 cycles
  Other Names: LoHP
  Arms: 1
Drug: Fluorouracil — Fluorouracil 400 mg/m2 infused over 10 min IV and Fluorouracil600 mg/m2 infused over 22 hours IV, Day 1 and 2 (De Grammont regimen)every 2 weeks for 12 cycles
  Other Names: 5-FU
  Arms: 2
Drug: Leucovorin — Leucovorin 200 mg/m2 infused over 1 hour IV on day 1 and day 2 (De Grammont regimen) every 2 weeks for 12 cycles
  Other Names: LV
  Arms: 2
Drug: Oxaliplatin — Oxaliplatin 85 mg/m2 as a 4 hour IV infusion, Day 1 every 4 weeks for 6 cycles
  Other Names: LoHP
  Arms: 2

SUMMARY:
This phase II trial will compare the efficacy and toxicity of the combination of Irinotecan and Oxaliplatin versus 5-FU/LV and Oxaliplatin as first line treatment in patients with locally advanced or metastatic gastric cancer

DETAILED DESCRIPTION:
There is no regimen considered standard in advanced gastric cancer. The reported response rates of 5-FU-based combination chemotherapy are higher than single agents (10-50%) but more toxic. The combination of 5-FU/LV and LOHP has demonstrated an ORR of 43%, median TTP of approximately 6,5 months and OS of 8,6 months in phase II trials, with an acceptable toxicity.

Irinotecan (CPT-11) is effective as salvage treatment in metastatic gastric cancer and has a synergistic activity with LOHP in preclinical trials

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic gastric cancer.
* Measurable or evaluable disease.
* Measurable disease is defined as at least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or 1 bidimensionally measurable lesion ≥ 20 X 10 mm. Lesions that are smaller or uni- or bidimensionally unmeasurable are considered as evaluable disease.
* Previous adjuvant chemotherapy with Irinotecan, Oxaliplatin and/or 5-FU based regimen. Patients who relapse within the first 6 months after the completion of adjuvant treatment are not eligible for the study.
* Karnofsky performance status > 70%.
* Age ≥18 years.
* Adequate liver (Bilirubin ≤ 1.5 UNL, SGOT/SGPT ≤ 4 UNL, ALP ≤ 2.5 UNL), renal (Creatinine ≤ 1.5 UNL) and bone marrow (ANC ≥ 1,500/mm3, PLT ≥ 100,000/mm3) function.
* Patients must be able to understand the nature of this study and give written informed consent.

Exclusion Criteria:

* Active infection
* History of serious cardiac disease (unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias)
* Previous radiotherapy within the last 4 weeks or > 25% of bone marrow.
* Patients with CNS metastases
* Patients with chronic diarrhea (at least for 3 months) or partial bowel obstruction.
* Malnutrition or loss of > 10% of body weight during the last month.
* Peripheral neuropathy ≥ grade 2
* Second primary malignancy, except for non-melanoma skin cancer and in situ cervical cancer.
* Psychiatric illness or social situation that would preclude study compliance.
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2004-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Objective Response Rates | Objective responses confirmed by CT or MRI (on 3rd and 6th cy)

SECONDARY OUTCOMES:
Time to progression | 1 year
Toxicity | Toxicity assessment on each chemotherapy cycle
Overall survival | 1 year
Quality of life | Assessment every two cycles
Symptoms improvement | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Boukovinas, MD, Principal Investigator — "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology
Locations (8):
- Greece (8):
  - University Hospital of Crete, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - State General Hospital of Larissa, Larissa
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus